CLINICAL TRIAL: NCT00699140
Title: Clinical Trial to Evaluate the Efficacy and the Safety of IGIV3I Grifols 10% (Human Intravenous Immunoglobulin) in Patients Diagnosed With Immune Thrombocytopenic Purpura
Brief Title: Clinical Trial in Patients Diagnosed With Immune Thrombocytopenic Purpura
Acronym: ITP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG202
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Immune (Idiopathic) Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 treatment group with IGIV3I Grifols (Experimental): Open label, non-randomized treatment group with IGIV3I Grifols
  Each patient received a total dose of 2 g/kg IGIV3I Grifols, given intravenously over either 2 days or 5 days in divided doses.
  Interventions: Biological: IGIV3I Grifols

INTERVENTIONS:
Biological: IGIV3I Grifols — Immune Globulin Intravenous (Human)
  Other Names: IGIV

SUMMARY:
The purpose of this study is to determine whether IGIV3I Grifols 10% is effective in the treatment of immune thrombocytopenic purpura.

DETAILED DESCRIPTION:
To determine if IGIV3I Grifols 10% is a consistently effective treatment in patients diagnosed with immune thrombocytopenic purpura with respect to:

1. Increase of platelet count ≥ 50x10^9/L (primary objective).
2. Time taken for the platelet count to reach ≥ 50x10^9/L.
3. The length of time the platelet count remains ≥ 50x10^9/L.
4. The maximum platelet level.
5. Regression of bleeding episodes during the first 10 or 14 days.

To determine if IGIV3I Grifols 10% is safe with respect to:

Nature, severity and frequency of adverse reactions during and after infusions by percentage of subjects and percentage of infusions.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged between 18 and 82 at the time of written consent.
2. Have confirmed diagnosis of chronic ITP and fulfil all the following criteria:

   * irrelevant history except for the symptoms of bleeding,
   * pattern of bleedings associated with platelet disorders,
   * physical examination irrelevant for the ITP, except for the signs of bleeding,
   * isolated thrombocytopenia in the blood count; apart from thrombocytopenia, the blood count is normal for the patient's age, or if abnormal, readily explained,
   * peripheral blood smear consistent with ITP: thrombocytopenia with platelets of normal size or slightly larger than normal, with absence of platelet clumps and giant platelets; normal red blood cell and white blood cell morphology,
   * confirmed diagnosis of immune thrombocytopenic purpura or, when any abnormal finding is present, additional diagnostic evaluation excludes other causes of thrombocytopenia.
   * Previous known diagnosis of ITP for at least 3 months.
3. To show a platelet count platelet count ≤ 20x10^9/L at the moment of the first infusion with the study product.
4. Have read the patient information and consent sheet, agreed to participate in the trial, and signed the consent sheet.
5. Be expected to receive treatment over 5 days and follow-up for 3 months.
6. For women of childbearing age, use adequate contraceptive method such as oral contraceptives, intrauterine device or tubal ligation during one-month period after the first infusion in the study.

Exclusion Criteria:

1. Have immune thrombocytopenia secondary to other pathologies or drug mediated thrombocytopenia.
2. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
3. Present important active bleeding due to other reasons apart from the ITP.
4. Exhibit an identifiable alternative cause of their thrombocytopenia, such as splenomegaly, family thrombocytopenia, bacteraemia, sepsis or active infection requiring or not therapy.
5. Are presenting renal dysfunction.
6. Have non-controlled arterial hypertension.
7. Have documented liver cirrhosis or any hepatic disorder with alanine aminotransferase (ALT) levels 2.5 times or more than the normal upper limit or bilirubin greater than 2 mg/dL.
8. Are presenting a cardiac disease including a history of coronary artery disease, angina pectoris or congestive heart failure.
9. Present known infection due to HIV or hepatitis C virus (HCV).
10. Have been previously treated with IVIG or anti-D immunoglobulin being unresponsive.
11. Have a history of serious adverse reactions or non-serious but frequent adverse reactions to intravenous immune globulin (IVIG) preparations or other products derived from blood.
12. Have known allergies to any IGIV3I Grifols components, such as D-sorbitol.
13. Are simultaneously participating in other clinical studies or have received an investigational drug in the 3 months prior to the start of the study.
14. Have been involved in the present study and being treated with the formulation at 5% (IGIV3I Grifols 5%).
15. Have conditions that might affect patient compliance.
16. Are unable to provide a storage serum sample just before the first dose of IGIV3I Grifols.
17. Are pregnant or nursing an infant child or unwilling to practice adequate birth control in 1-month period after the first infusion in the study.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: María Teresa Álvarez, MD, Principal Investigator — Hospital General Universitario La Paz
Locations (7):
- Russia (2):
  - Federal Research Clinical Centre of Pediatric Hematology, Oncology and Immunology Roszdrava, Moscow
  - Haematology Research Centre of Russian Academy of Medical Science, Moscow
- Spain (4):
  - Hospital General Vall d´Hebron, Barcelona
  - . Hospital de León, León
  - Hospital General Universitario La Paz, Madrid
  - Hospital Universitario La Fe, Valencia
- Hillingdon Hospital, Middlesex, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Treatment Group With IGIV3I: Open label, non-randomized treatment group with IGIV3I Grifols
  IGIV3I Grifols: Immune Globulin Intravenous (Human)
  Each patient received a total dose of 2 g/kg IGIV3I Grifols, given intravenously over either 2 days or 5 days in divided doses
Period: Overall Study
Arm/Group | 1 Treatment Group With IGIV3I
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 1 Treatment Group With IGIV3I
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 43 [20 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 12
  United Kingdom | 2
  Spain | 4
Subjects with medical history of splenectomy [Number; unit: participants]
  Yes | 9
  No | 9
Subjects with haemorrhagic history [Number; unit: participants]
  Yes | 13
  No | 5
Platelet count [Median (Full Range); unit: platelets x 10^-9/L] | 8.5 [3.0 to 36.0]

OUTCOME MEASURES:

1. Primary Outcome: Responder Patients
Description: The primary efficacy endpoint was the proportion of patients who reached a platelet count ≥ 50x10^9/L.
Time Frame: At any time during the study period (The platelet count was measured at Days 1-6, 10, 14. 21, 30, 60, 90).
Population: All 18 subjects received at least one infusion (at any dose) of IGIV3I Grifols and were included in the intent-to-treat (ITT) population for efficacy and safety analysis.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 1 Treatment Group With IGIV3I
Number analyzed (Participants) | 18
percentage of subjects | 72.2 [50.2 to 88.4]

2. Secondary Outcome: Maximum Platelet Level Reached During the Follow-up Period
Description: Platelet count was measured at various time points in the follow-up period after infusion.
Time Frame: During the follow-up period (time points: Days 6, 10, 14, 21, 30, 60, 90 post-first infusion day [Day 1])
Population: The maximum platelet counts were taken from the population who responded to treatment (platelet count ≥ 50x10^9/L). If any patient received banned medication due to ITP progression during the study, the values obtained after patients received treatment were excluded.
Measure: Median (Full Range); unit: platelets x 10^-9/L
Arm/Group | 1 Treatment Group With IGIV3I
Number analyzed (Participants) | 13
platelets x 10^-9/L | 146.0 [71.0 to 763.0]

3. Secondary Outcome: Time to Reach Platelet Count ≥ 50x10^9/L (≤ Days)
Description: The time taken for the platelet count to reach ≥ 50x10^9/L from first dose
Time Frame: At any time during the study period (time points: Days 1-6, 10, 14, 21, 30, 60, 90 post-first infusion day [Day 1])
Population: From all 18 subjects who received at least one infusion and were included in the intent-to-treat (ITT) population but only 13 responded to the treatment
Measure: Median (Full Range); unit: days
Arm/Group | 1 Treatment Group With IGIV3I
Number analyzed (Participants) | 13
days | 2 [0 to 5]

4. Secondary Outcome: Length of Time Platelet Count Remains ≥ 50x10^9/L (≥ Days)
Description: Length of time platelet count remained ≥ 50x10^9/L from first dose (Day 1)
Time Frame: At any time during the study period (up to 3 months [90 days])
Population: From all 18 subjects who received at least one infusion and were included in the intent-to-treat (ITT) population only 13 responded to the treatment
Measure: Median (Full Range); unit: days
Arm/Group | 1 Treatment Group With IGIV3I
Number analyzed (Participants) | 13
days | 9 [3 to 61]

5. Secondary Outcome: Regression of Hemorrhages.
Description: Percentage of subjects with regression of hemorrhages of Types 1 to 3:
  * Type 0: Patients without symptoms of bleeding at the first infusion continue without presenting spontaneous bleeding
  * Type 1: Patients with bleeding symptoms at the first infusion had a reduction of the size of large ecchymoses, and no spontaneous appearance of new ecchymoses
  * Type 2: Patients with bleeding symptoms at the first infusion had a decrease in the number of cutaneous petechiae, or the extent of the affected area of the body decreased
  * Type 3: Patients had active mucosal bleedings at the first infusion, these episodes stopped without re-bleeding, and there was no occurrence of new spontaneous mucosal hemorrhages (e.g., gingival bleeding, epistaxis)
Time Frame: First 10 to14 days since the first infusion day (Day 1)
Population: ITT population: patients who received at least one infusion of the study drug
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 1 Treatment Group With IGIV3I
Number analyzed (Participants) | 18
percentage of subjects | 83.3 [62.3 to 95.3]

6. Secondary Outcome: Frequency of Adverse Reactions During and After Infusions by Percentage of Patients
Description: All adverse events (AEs) are tabulated and summarized. The incidence, severity, and causal relationship of the AEs to IGIV3I Grifols are presented by system organ class after medical coding according to the version 15.0 of Medical Dictionary for Regulatory Activities (MedDRA). The frequency of patients with at least one AE and adverse drug reactions are estimated.
Time Frame: At any time during the study period (from patient's signature of the informed consent form until 3 months of follow-up)
Population: ITT population: patient who received one infusion with the study drug.
Measure: Number; unit: percentage of patients
Groups:
- 1 Treatment Group With IGIV3I: Open label, non-randomized treatment group with IGIV3I Grifols. IGIV3I Grifols: Immune Globulin Intravenous (Human). All adverse events (AEs) are tabulated and summarized. Incidence, severity, and causal relationship of the AEs to IGIV3I Grifols are presented by system organ class after medical coding according to the version 15.0 of MedDRA.
  The frequency of patients and infusions associated with at least one AE are estimated as the primary safety endpoint.
Arm/Group | 1 Treatment Group With IGIV3I
Number analyzed (Participants) | 18
percentage of patients
  Frequency of patients with AEs | 88.9
  Frequency of patients with adverse drug reactions | 38.9

7. Secondary Outcome: Frequency of Adverse Reactions During and After Infusions by Percentage of Infusions
Description: All adverse events (AEs) are tabulated and summarized. The incidence, severity, and causal relationship of the AEs to IGIV3I Grifols are presented by system organ class after medical coding according to the version 15.0 of Medical Dictionary for Regulatory Activities (MedDRA). The frequency of infusions associated with at least one AE and adverse drug reactions are estimated.
Time Frame: At any time during the study period (from patient's signature of the informed consent form until 3 months of follow-up)
Population: ITT population: patient who received at least one infusion with the study drug.
Measure: Number; unit: percentage of infusions
Groups:
- 1 Treatment Group With IGIV3I Grifols: Open label, non-randomized treatment group with IGIV3I Grifols
  IGIV3I Grifols: Immune Globulin Intravenous (Human)
  Each patient received a total dose of 2 g/kg IGIV3I Grifols, given intravenously over either 2 days or 5 days in divided doses.
Arm/Group | 1 Treatment Group With IGIV3I Grifols
Number analyzed (Participants) | 18
percentage of infusions
  Frequency of infusions with adverse events | 26.3
  Frequency of infusions with adverse drug reactions | 24.6

8. Secondary Outcome: Changes in Vital Signs and Clinically Relevant Changes in Laboratory Parameters After the Infusions, Including Renal Function (Creatinine Levels)
Description: Laboratory parameters at each treatment day and visit are summarized by patient. Results were marked as normal/abnormal (whether the result is below, within or above the respective reference range) and relevant/irrelevant (as determined by the investigator). The number of abnormal values considered clinically relevant changes (based on the investigator's judgment) was listed.
Time Frame: At any time during the study period (from patient's signature of the informed consent form until 3 months of follow-up)
Population: Intent-to-treat population
Measure: Number; unit: participants
Groups:
- 1 Treatment Group With IGIV3I Grifols: Open label, non-randomized treatment group with IGIV3I Grifols
  Each patient received a total dose of 2 g/kg IGIV3I Grifols, given intravenously over either 2 days or 5 days in divided doses.
  IGIV3I Grifols: Immune Globulin Intravenous (Human)
Arm/Group | 1 Treatment Group With IGIV3I Grifols
Number analyzed (Participants) | 18
participants
  Clinically relevant changes in vital signs | 0
  Clinically relevant changes in lab parameters | 7

9. Secondary Outcome: Viral Safety Through the Investigation of Patients Virology Status (Hepatitis A Virus [HA
Description: The results of HIV-1 and -2 antibodies, HCV antibody, HBsAg, HBV antibodies, HAV antibodies, HIV nucleic acid amplification test [NAT], and HCV NAT on Day 1, Day 14, and at Month 1, Month 2 and Month 3 were recorded for several of these markers (as appropriate). A comparison of negative viral markers on Day 1 and Month 3 was performed
Time Frame: At any time during the study period (from patient's signature of the informed consent form until 3 months of follow-up)
Population: Intent-to-treat population
Measure: Number; unit: seroconversions
Arm/Group | 1 Treatment Group With IGIV3I
Number analyzed (Participants) | 18
seroconversions | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: At any time during the study period (from patient´s signature of the informed consent until 3 months of follow-up)
Groups:
- 1 Treatment Group With IGIV3I Grifols: Open label, non-randomized treatment group with IGIV3I Grifols
  IGIV3I Grifols: Immune Globulin Intravenous (Human)
Arm/Group | 1 Treatment Group With IGIV3I Grifols
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Treatment Group With IGIV3I Grifols (N=18)
Thrombosis (Vascular disorders) | 1 (1) — A male subject of 54-year-old, with morbid obesity, sedentary lifestyle, previous steroid treatment and difficulty with line insertion was diagnosed with deep venous thrombosis and hospitalized. The subject recovered from the event.
Haemoglobin decreased (Investigations) | 1 (1) — A 75-year-old male with high blood glucose levels and hypertension presented a drop in hemoglobin from 11.7 g/dL to 9.8 g/dL. The reaction was transient with no complications or clinical symptoms of hemolysis. The subject was recovered from the event
Leukopenia (Blood and lymphatic system disorders) | 1 (1) — A 75-year-old male with high blood glucose levels and hypertension presented a drop in leukocyte count from 5.3x10^9/L to 2.7x10^9/L. The reaction was transient, with no complications. The subject was discharged from hospital totally recovered
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Treatment Group With IGIV3I Grifols (N=18)
Petechiae (Skin and subcutaneous tissue disorders) | 12 (15) — All of these events were considered not related to the study drug
Ecchymosis (Skin and subcutaneous tissue disorders) | 8 (11) — Only 1 out of 11 events was considered related to the study drug
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) — It was considered related to the study drug
Rash (Skin and subcutaneous tissue disorders) | 2 (2) — Only 1 of the 2 events was considered related to the study drug
Pyrexia (General disorders) | 4 (4) — Three out of 4 events were considered related to the study drug
Chills (General disorders) | 2 (2) — All of 2 events were considered related to the study drug
Fatigue (General disorders) | 1 (2) — Two events were considered related to the study drug
Abdominal distension (Gastrointestinal disorders) | 1 (3) — One patient had 3 events that were considered not related to the study drug
Gingival bleeding (Gastrointestinal disorders) | 2 (2) — Two patients had 2 events that were considered not related to the study drug
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (2) — A patient had 2 events that were considered not related to the study drug
Nausea (Gastrointestinal disorders) | 1 (1) — It was considered related to the study drug
Vomiting (Gastrointestinal disorders) | 1 (1) — It was considered related to the stuy drug
Headache (Nervous system disorders) | 7 (15) — Twelve out of 15 events were considered related to the study drug
Radicular syndrome (Nervous system disorders) | 1 (1) — It was considered related to the study drug
Haematoma (Vascular disorders) | 1 (1) — It was considered not related to the study drug
Hypertension (Vascular disorders) | 2 (3) — Two patients had 3 events that were considered related to the study drug
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) — A patient had 2 events that were considered not related to the study drug
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — It was considered not related to the study drug
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — A patient had 1 event that was considered not related to the study drug
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (2) — A patient had 2 events that were considered related to the study drug
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) — A patient had 1 event that was considered not related to the study drug
Alanine aminotransferase increased (Investigations) | 1 (1) — It was considered not related to the study drug
Blood cholesterol increased (Investigations) | 1 (1) — It was considered not related to the study drug
Blood triglycerides increased (Investigations) | 1 (1) — It was considered not related to the study drug
Lipids abnormal (Investigations) | 1 (1) — It was considered not related to the study drug
Drug hypersensitivity (Immune system disorders) | 1 (1) — It was considered related to the study drug
Nasopharyngitis (Infections and infestations) | 1 (2) — A patient had 2 events that were considered not related to the study drug
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) — It was considered related to the study drug
Haematuria (Renal and urinary disorders) | 1 (1) — It was considered not related to the study drug

LIMITATIONS AND CAVEATS:
The patient number was based on European Medicines Agency guidance to evaluate IVIG products in ITP patients (EMEA/CPMP/BPWG/388/95 rev.1, June 2000, in force when the study was designed): at least 15 subjects were sufficient for the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No